CLINICAL TRIAL: NCT00003434
Title: A Pilot Study of Active Immunotherapy With Carcinoembryonic Antigen Peptide-Pulsed, Autologous Human Cultured Dendritic Cells in Patients With Resected, Stage I, II and III Pancreatic Adenocarcinoma Expressing Carcinoembryonic Antigen
Brief Title: Biological Therapy in Stage I, Stage II, or Stage III Surgically Resected Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1259; DUMC-97093; NCI-G98-1457; CDR0000066460 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-04-27 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Pancreatic Cancer
Keywords: stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — CAP1-6D; Hepatitis B Surface Antigens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: carcinoembryonic antigen peptide 1
Biological: hepatitis B antigen peptide

SUMMARY:
Rational: White blood cells that have been treated with carcinoembryonic antigen peptide-1 may help the body build an immune response to and kill tumor cells that express CEA.

Purpose: Phase II trial to study the effectiveness of white blood cells plus carcinoembryonic antigen peptide-1 in treating patients with stage I, stage II, or stage III pancreatic cancer that has been surgically removed.

DETAILED DESCRIPTION:
Objective: I. Perform a pilot study of active immunotherapy with autologous dendritic cells pulsed with the CEA peptide, CAP-1, after surgical resection in patients with CEA expressing pancreatic cancer. II. Perform laboratory analysis to monitor the presence, persistence, and function of CAP-1 specific T-cells in this patient population.

Outline: Patients undergo leukapheresis for up to 4.5 hours prior to vaccination. Half of the collected dendritic cells are pulsed with carcinoembryonic antigen (CEA) peptide and the other half are pulsed with hepatitis B antigen peptide (HBsAg). Equal doses of CEA and HBsAg peptide pulsed dendritic cells are administered intravenously over 3 minutes every 4 weeks for a total of 6 doses each. Patients undergo a second leukopheresis 2 weeks after the last dose of immunotherapy to obtain specimens for immunologic tests. Patients are followed at weeks 22, 36, 48, and every 6 months thereafter.

Project Accrual: A total of 24 patients will be accrued for this study over 2 years.

ELIGIBILITY:
Disease Characteristics:

* Histologically confirmed stage I, II, or III adenocarcinoma of the pancreas Resected with no gross residual disease At least 50% of tumor cells must be CEA positive and stain with at least moderate intensity HLA-A2 positive

Patient Characteristics:

* Age: 18 and over
* Performance status: Karnofsky 70-100%
* Life expectancy: Greater than 6 months
* Hematopoietic: Absolute neutrophil count at least 1000/mm3
* Hepatic: Bilirubin less than 2.0 mg/dL SGOT and alkaline phosphatase less than 4 times the upper limit of normal No hepatic failure
* Renal: Creatinine less than 2.0 mg/dL OR Creatinine clearance greater than 50 mL/min
* Cardiovascular: No New York Heart Association class III or IV heart disease
* Pulmonary: No concurrent asthma or chronic obstructive pulmonary disease

Other:

* No other malignancy except nonmelanoma skin cancer or controlled superficial bladder cancer within the past 5 years.
* No history of autoimmune diseases such as inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, rheumatoid arthritis, or multiple sclerosis
* No active acute or chronic infection such as urinary tract infection, HIV, or viral hepatitis
* No active infectious enteritis or eosinophilic enteritis Not pregnant or nursing Fertile patients must use effective contraception

Prior Therapy:

* Biologic therapy: At least 4 weeks since immunotherapy. No other concurrent immunotherapy
* Chemotherapy: At least 4 weeks since chemotherapy and recovered. No concurrent chemotherapy
* Endocrine therapy: No concurrent corticosteroid or immunosuppressive therapy. At least 6 weeks since steroid therapy
* Radiotherapy: At least 4 weeks since radiotherapy and recovered
* Surgery: Recovered from prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 1998-06; Primary Completion 2002-08 (Actual); Study Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Morse, MD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States